CLINICAL TRIAL: NCT05123599
Title: A Phase 1b, Open-label, Single-arm, Multicenter Study to Assess Efficacy, Safety, and Tolerability of Treatment With JNJ-73763989, JNJ-64300535, and Nucleos(t)Ide Analogs in Virologically Suppressed, HBeAg-negative Participants With Chronic Hepatitis B Virus Infection
Brief Title: A Study of JNJ-73763989, JNJ-64300535, and Nucleos(t)Ide Analogs in Virologically Suppressed, Hepatitis B e Antigen (HBeAg)- Negative Participants With Chronic Hepatitis B Virus Infection
Acronym: OSPREY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR109042; 2020-005584-30 (EudraCT Number); 73763989PAHPB1006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-11-16; First posted 2021-11-17 (Actual); Last update posted 2025-05-26 (Actual); Status verified 2025-05

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JNJ-73763989 plus JNJ-64300535 plus Nucleos(t)ide Analogs (NAs) (Experimental): Participants will receive JNJ-73763989 subcutaneous (SC) injection once every 4 weeks (q4w), NA (either Entecavir monohydrate [ETV], Tenofovir disoproxil or Tenofovir alafemide [TAF]) oral tablets once daily (qd) and JNJ-64300535 intramuscular (IM) injection q4w. From day 187, participants will receive treatment with NA oral tablets qd up to Week 36.
  Interventions: Drug: JNJ-73763989; Biological: JNJ-64300535; Drug: ETV monohydrate; Drug: Tenofovir disoproxil; Drug: TAF

INTERVENTIONS:
Drug: JNJ-73763989 — JNJ-73763989 injection will be administered subcutaneously.
  Other Names: JNJ-3989
Biological: JNJ-64300535 — JNJ-64300535 deoxyribonucleic acid (DNA) vaccine injection will be administered intramuscularly.
  Other Names: JNJ-0535
Drug: ETV monohydrate — ETV monohydrate film-coated tablets will be administered orally.
Drug: Tenofovir disoproxil — Tenofovir disoproxil film-coated tablets will be administered orally.
Drug: TAF — TAF film-coated tablets will be administered orally.

SUMMARY:
The purpose of this study is to evaluate the efficacy of the study intervention based on hepatitis B surface antigen (HBsAg) levels.

DETAILED DESCRIPTION:
JNJ-73763989 is a liver-targeted antiviral therapeutic for subcutaneous injection designed to treat chronic hepatitis B virus (HBV) infection via a ribonucleic acid interference (RNAi) mechanism. JNJ-64300535 is a DNA vaccine encoding the core protein and the Polymerase (Pol) protein of HBV. The therapeutic vaccine aims at inducing T-cell-specific immunity against HBV antigens in participants with chronic hepatitis B (CHB). Selected nucleos(t)ide analogs (NAs) used in this study are approved treatments of chronic HBV infection. This study is designed to assess efficacy, safety, and tolerability of a 24-week (Day 1 to Week 24) combination treatment with JNJ-73763989 + NA + JNJ-64300535. The study consists of a Screening phase (4 weeks), Treatment period with JNJ-73763989, NA and JNJ-64300535 (187 days), and a follow-up period (FU Week 1 till FO Week 48). Safety will be assessed by adverse events (AEs), clinical safety laboratory assessments, electrocardiograms (ECGs), vital signs and physical examinations. The total duration of the study is up to 88 weeks (including 4 weeks of screening).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be medically stable based on physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening. Any abnormalities, must be consistent with the underlying illness in the study population and this determination must be recorded in the participant's source documents and initialed by the investigator
* Participants must have a body mass index (BMI; weight in kilograms [kg] divided by the square of height in meters) between 19.0 and 32.0 kilograms per meter square (kg/m^2), extremes included
* A woman of childbearing potential must have a negative highly sensitive serum pregnancy test (beta-human chorionic gonadotropin) at screening and a negative urine pregnancy test on Day 1 before the first dose of study intervention
* Participants must have chronic hepatitis B virus (HBV) infection. HBV infection must be documented by serum hepatitis B surface antigen (HBsAg) positivity at screening. In addition, chronicity must be documented by any of the following, at least 6 months prior to screening: serum HBsAg positivity, hepatitis B e antigen (HBeAg) positivity or HBV deoxyribonucleic acid (DNA) positivity, alanine aminotransferase (ALT) elevation above upper limit of normal (ULN) without another cause than HBV infection, documented transmission event. If none of the above are available, the following ways of documenting chronicity are acceptable at the time of screening: liver biopsy with changes consistent with chronic HBV, or absence of marker for acute HBV infection such as positive immunoglobulin M (IgM) anti- hepatitis B surface protein (HBs) and anti- hepatitis B core protein (HBc) antibodies. Virologically suppressed participants should: a) be HBeAg-negative and anti- hepatitis B e (HBe) positive, b) be on stable HBV treatment, defined as currently receiving nucleos(t)ide analog (NA) treatment for at least 6 months prior to screening and having been on the same NA treatment regimen (at the same dose) as used in this study for at least 3 months at the time of screening, c) have serum HBV deoxyribonucleic acid (DNA) less than (<) 60 International units per milliliter (IU/mL) on 2 sequential measurements at least 6 months apart (one of which is at screening), and d) have documented ALT values <2.0* ULN on 2 sequential measurements at least 6 months apart (one of which is at screening)
* Participants must have: a) Fibroscan liver stiffness measurement less than or equal to (<=) 9.0 kPa within 6 months prior to screening or at the time of screening, or b) If a Fibroscan result is not available: a liver biopsy result classified as Metavir F0-F2 within 1 year prior to screening

Exclusion Criteria:

* History or evidence of clinical signs or symptoms of hepatic decompensation, including but not limited to: portal hypertension, ascites, hepatic encephalopathy, esophageal varices
* Participants with a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which are considered cured with minimal risk of recurrence)
* Participants with any history of or current clinically significant skin disease requiring regular or periodic treatment
* Participants with clinically relevant alcohol or drug abuse within 12 months of screening
* Participants who had major surgery (example, requiring general anesthesia), excluding diagnostic surgery, within 12 weeks before screening; or will not have fully recovered from surgery; or have surgery planned during the time of expected participation in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a Reduction of at Least 2 log10 International Units per Milliliter (IU/mL) in Hepatitis B Surface Antigen (HBsAg) Levels from Baseline to Week 36 | Baseline to Week 36 (end of study intervention)
  Percentage of participants with a reduction of at least 2 log10 IU/mL in HBsAg levels from baseline to Week 36 will be reported.

SECONDARY OUTCOMES:
Percentage of Participants with at Least 3-fold Increase in Hepatitis B Virus (HBV)- Specific T-Cell Response Against Vaccine Antigen HBV Core and/or Pol | From Day 103 up to Week 84
  Percentage of participants with at least 3-fold increase in HBV-specific T-cell response against vaccine antigen HBV core and/or pol as assessed by enzyme-linked immunospot (ELISpot) will be reported.
Percentage of Responders Against Vaccine Antigen HBV Core and/or Pol | Week 28
  Percentage of responders against vaccine antigen HBV core and/or Pol as assessed by ELISpot will be reported. A responder is defined as a participant with at least a 3-fold increase in HBV-specific T-cell response from the start of vaccination against the vaccine antigen core and/or pol, at least at the last timepoint during the vaccination period.
Percentage of Participants with Adverse Events (AEs) | Up to Week 84
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Percentage of Participants with Serious AEs | Up to Week 84
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Percentage of Participants with Abnormalities in Clinical Laboratory Tests | Up to Week 84
  Percentage of participants with abnormalities in clinical laboratory tests (hematology, blood biochemistry, blood coagulation, urinalysis, urine chemistry, and renal biomarkers) will be reported.
Percentage of Participants with Abnormalities in 12- lead Electrocardiograms (ECGs) | Up to Week 84
  Percentage of participants with abnormalities in 12- lead ECGs will be reported.
Percentage of Participants with Abnormalities in Vital Signs | Up to Week 84
  Percentage of participants with abnormalities in vital signs will be reported.
Percentage of Participants with Abnormalities in Physical Examinations | Up to Week 84
  Percentage of participants with abnormalities in physical examinations will be reported.
Percentage of Participants with Solicited Local AEs for JNJ-64300535 up to 7 Days Post Each Vaccination | 7 days post each vaccination (Up to Day 194)
  Solicited local AEs include (injection site pain/tenderness, erythema and swelling at the study vaccine injection site and the extent (largest diameter) of any erythema and swelling [using the ruler supplied]) will be reported after 7 days of each vaccination.
Percentage of Participants with Solicited Systematic AEs for JNJ-64300535 up to 7 Days Post Each Vaccination | 7 days post each vaccination (Up to Day 194)
  Solicited systemic AEs (include body temperature, fatigue, headache, nausea, myalgia) will be reported after 7 days of each vaccination.
Change from Baseline Over Time in HBsAg Levels | Baseline up to Week 84
  Change from baseline over time in HBsAg levels will be reported.
Change from Start of Vaccination Over Time in HBsAg Levels | From Day 103 up to Week 84
  Change from start of vaccination over time in HBsAg levels will be reported.
Percentage of Participants with HBsAg, HBV Deoxyribonucleic Acid (DNA) and Alanine Aminotransferase (ALT) Levels Below/Above Different Cut-offs | Up to Week 84
  Percentage of participants with HBsAg, HBV DNA and ALT levels below/above different cut-offs will be reported.
Percentage of Participants with HBsAg Seroclearance | Up to Week 84
  Percentage of participants with HBsAg seroclearance (HBsAg negativity) will be reported.
Percentage of Participants with HBsAg Seroconversion | Up to Week 84
  Percentage of participants with HBsAg seroconversion (HBsAg negativity and anti-HBs antibody positivity) will be reported.
Time to Achieve HBsAg Seroclearance | Up to Week 84
  Time to achieve HBsAg seroclearance will be reported.
Time to Achieve HBsAg Seroconversion | Up to Week 84
  Time to achieve HBsAg seroconversion will be reported.
Percentage of Participants Meeting Nucleos(t)ide Analog (NA) Treatment Completion Criteria | Week 38 and Week 40
  Percentage of participants meeting NA treatment completion criteria will be reported.
Percentage of Participants with Virological Breakthrough | Up to Week 36
  Percentage of participants with virological breakthrough (confirmed on-treatment HBV DNA increase by greater than [>] 1 log10 IU/mL from nadir or confirmed on-treatment HBV DNA level >200 IU/mL in participants who had HBV DNA level less than [<] lower limit of quantification [LLOQ] of the HBV DNA assay) will be reported.
Percentage of Participants with HBsAg Seroclearance at Week 60 and Week 84 | Weeks 60 and 84
  Percentage of participants with HBsAg seroclearance at Weeks 60 and 84 (during follow-up period) will be reported.
Percentage of Participants with HBV DNA <LLOQ at Week 60 and Week 84 | Weeks 60 and 84
  Percentage of participants with HBV DNA <LLOQ at Weeks 60 and 84 (during follow-up period) will be reported.
Percentage of Participants with Viral Flares | From Week 36 to Week 84
  Percentage of participants with viral flares will be reported.
Percentage of Participants with Biochemical Flares | From Week 36 to Week 84
  Percentage of participants with biochemical flares will be reported.
Number of TriGrid Delivery System (TDS)-Intramuscular (IM) version 2.0 Device Fault Conditions by Type | From Day 103 to Day 187
  Number of TDS-IM v2.0 device fault conditions by type will be observed. User reported fault conditions will be documented to enable assessment of the device reliability. Device functions to be assessed include electrode/needle deployment, JNJ-64300535 administration, and electroporation application.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- Belgium (2):
  - UZ Antwerpen, Edegem
  - UZA-SGS, Edegem
- France (2):
  - Hopital Beaujon, Clichy
  - Hopital de La Croix Rousse, Lyon
- Italy (2):
  - Irccs Ospedale Maggiore Di Milano, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- New Zealand Clinical Research, Auckland, New Zealand
- ID Clinic, Mysłowice, Poland
- Spain (2):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. Marques de Valdecilla, Santander
- Taiwan (2):
  - E-DA Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan District
- Kings College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency